CLINICAL TRIAL: NCT02378272
Title: RCT on Care Manager Organization for Management of Mild-moderate Depression in the Primary Care Setting, Sweden
Brief Title: Care Manager - Coordinating Care for Person Centered Management of Depression in Primary Care
Acronym: PRIM-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS 1938-2013
Record Dates: First submitted 2015-02-02; First posted 2015-03-04 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: Care Manager; Primary Care; Depressive symptoms; quality of life; return to work
MeSH Terms: conditions — Depression | interventions — Case Managers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care manager for depression (Experimental): A district nurse will apply around 15-25% of working time as care coordinator (care manager for depression) at PCC for management of care for all recruited patients with depression
  Interventions: Other: care manager for depression
- Treatment As Usual (No Intervention): Management of recruited patients with depression continued as usually applied at PCC

INTERVENTIONS:
Other: care manager for depression — District nurse (care manager for depression) providing clinical services ( in cooperation with GP) as patient information and education on patient's preferred treatment, development of care plan, assessment of patient's depressive symptoms and regular telephone contacts.
  Arms: Care manager for depression

SUMMARY:
The aim of the project is to explore if a complementary addition of a care manager for depression treatment in the primary care setting has positive effects concerning reduction of the patients' depressive symptoms as well as improvement of daily function and quality of life in a short- and long-term perspective compared with the traditional Swedish primary care organization. The aim is also to evaluate the care manager function in a health economic perspective.

The specific aims are to develop and evaluate an evidence-based care manager program for patients with mild to moderate depression and to compare the evidence-based care manager program to treatment as usual (TAU) in terms of their short- and long-term effects on symptom remission, treatment adherence, care satisfaction, and self-efficacy as well as to perform a cost - effectiveness analysis of the care manager program, i.e. to evaluate the effects of the program on patients' health in relation to the running costs of the program.

DETAILED DESCRIPTION:
Methods The research questions will be tested in a randomised controlled trial with follow ups 3 and 6 months in the primary care setting in cooperation between universities of Gothenburg, Karolinska Institute and primary care centres (PCC) of regions/county councils of Västra Götaland, and Dalarna.

Design A cluster randomized controlled trial of two groups (intervention and control). Randomization will be at the level of the primary care centers (PCCs).

Population of study Patients aged 18 and up that visit one of 20 different urban and rural PCCs.

Randomization All PCCs in the participating regions without employed onsite mental health professionals are invited to participate in the study. Around twenty practices will be matched into 10 blocks by depression treatment practices, thereafter 1 practice from each block will be randomly assigned to receive the care manager intervention program.

Intervention At the intervention practices, a district nurse will apply around 15-25% of working time as care coordinator for management of care for the patients with depression. Before patient recruitment begins, physicians and the nurse/district nurse (care manager) will participate in sessions for training in providing clinical services (patient information and education on patient's preferred treatment, assessment of patient's depressive symptoms and regular telephone contacts, follow up visits etc).

Recruitment of patients and Data collection Patients aged 18 and up that visit primary health care centres and are diagnosed by the General Practitioner (GP) with light/medium depression disorder according to PRIME-MD (4). The patients will be monitored up to 6 months after inclusion in the study by an individual interview (first visit, 3 and 6 months).

All parameters will be assessed at baseline and 3 and 6 months; prescription of antidepressants, number of days of labour lost, socio-demographic and economic variables, alcohol consumption, physical activity, and ethnicity. BDI-II, EuroQoL-5D, Work Ability Instrument (WAI) Karasek Job strain Model , medication, other treatment (psychological, counselling, or other).

For somatic health reasons, also blood pressure and p-glucose will be monitored, and blood samples for bio-bank storage.

Outcome criteria Change in: depression symptoms (BDI-II), work ability index (WAI), Job strain (Karasek), EQ-5D, QALYs from baseline to 3 and 6 months. Amount of sick listing (days, %), days of labour lost.

Statistical analysis Analysis of covariance, controlling for baseline value, will be used to estimate the overall treatment effectiveness (difference in score) at final follow-up. Subgroup analysis by gender as well as age adjustments will also be performed.

Power calculation The primary variable is the level of depression (as measured by the BDI-II) and analyzed in an ANCOVA model with repeated measures. In order to detect an effect of 3 units in the difference between the two groups, with a power of 80% and a significance level of 10% (two-sided) about 200 patients is needed in each group (9). The underlying assumption is a standard deviation in the group of 10 units, a within-subject correlation of 0.4, and a within-cluster-correlation of 0.1, i.e. a design effect of 1.9 to correct for having a cluster analysis.

Cost-effectiveness analysis A cost- effectiveness analysis (CEA) with quality-adjusted life years (QALY) as measure of effect will be performed.

The region Västra Götaland has proclaimed interest in the study, and financially supports the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed mild-moderate depression,
* 18 - 80 years,
* attending primary care center

Exclusion Criteria:

* schizophrenia,
* abuse/addiction,
* psychosis,
* bipolar syndrome,
* suicidal ideation or earlier suicide attempt,
* ongoing deep depression,
* generalized anxiety syndrome,
* not communicable in Swedish

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of level of depression (Self-reported level of depressive symptoms measured by Beck Depression Inventory II) | 0- 6 months
  Self-reported level of depressive symptoms measured by Beck Depression Inventory II

SECONDARY OUTCOMES:
Sick-listing (Amount of sick-listing days during 0-6 months observation period) | 6 months
  Amount of sick-listing days during 0-6 months observation period
Change of level of job strain (Perception of job strain measured by Karasek Job Strain Model) | 0-6 months
  Perception of job strain measured by Karasek Job Strain Model
Change of level of Quality of Life (Self-reported level of perceived Quality of Life measured by EQ-5D) | 0- 6 months
  Self-reported level of perceived Quality of Life measured by EQ-5D
Change of level of Work Ability (Self-reported level of perceived work ability measured by Work Ability Index) | 0 - 6 months
  Self-reported level of perceived work ability measured by Work Ability Index

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Björkelund, Principal Investigator — Göteborg University
Locations (1):
- Department of Primary Health Care, Sahlgrenska Academy, Gothenburg, Region Västra Götaland, Sweden

REFERENCES:
- [Result] Bjorkelund C, Svenningsson I, Hange D, Udo C, Petersson EL, Ariai N, Nejati S, Wessman C, Wikberg C, Andre M, Wallin L, Westman J. Clinical effectiveness of care managers in collaborative care for patients with depression in Swedish primary health care: a pragmatic cluster randomized controlled trial. BMC Fam Pract. 2018 Feb 9;19(1):28. doi: 10.1186/s12875-018-0711-z. PMID 29426288
- [Result] Holst A, Ginter A, Bjorkelund C, Hange D, Petersson EL, Svenningsson I, Westman J, Andre M, Wikberg C, Wallin L, Moller C, Svensson M. Cost-effectiveness of a care manager collaborative care programme for patients with depression in primary care: economic evaluation of a pragmatic randomised controlled study. BMJ Open. 2018 Nov 12;8(11):e024741. doi: 10.1136/bmjopen-2018-024741. PMID 30420353
- [Result] Petersson EL, Hange D, Udo C, Bjorkelund C, Svenningsson I. Long-term effect of a care manager on work ability for patients with depression - the PRIM-CARE RCT. Work. 2022;72(2):601-609. doi: 10.3233/WOR-205272. PMID 35527596
- [Result] Holst A, Labori F, Bjorkelund C, Hange D, Svenningsson I, Petersson EL, Westman J, Moller C, Svensson M. Cost-effectiveness of a care manager collaborative care programme for patients with depression in primary care: 12-month economic evaluation of a pragmatic randomised controlled trial. Cost Eff Resour Alloc. 2021 Aug 17;19(1):52. doi: 10.1186/s12962-021-00304-5. PMID 34404426
- [Result] Af Winklerfelt Hammarberg S, Bjorkelund C, Nejati S, Magnil M, Hange D, Svenningsson I, Petersson EL, Andre M, Udo C, Ariai N, Wallin L, Wikberg C, Westman J. Clinical effectiveness of care managers in collaborative primary health care for patients with depression: 12- and 24-month follow-up of a pragmatic cluster randomized controlled trial. BMC Prim Care. 2022 Aug 9;23(1):198. doi: 10.1186/s12875-022-01803-x. PMID 35945493
- [Derived] Augustsson P, Petersson EL, Bjorkelund C, Persson Kylen S, Wikberg C. Organisational and social work-environment experiences after care manager implementation: a repeated cross-sectional study in Swedish primary care. Scand J Prim Health Care. 2025 Jul 28:1-12. doi: 10.1080/02813432.2025.2538486. Online ahead of print. PMID 40726123
- [Derived] Svenningsson I, Hange D, Udo C, Tornbom K, Bjorkelund C, Petersson EL. The care manager meeting the patients' unique needs using the care manager model-A qualitative study of experienced care managers. BMC Fam Pract. 2021 Sep 3;22(1):175. doi: 10.1186/s12875-021-01523-8. PMID 34474682
- [Derived] Svenningsson I, Petersson EL, Udo C, Westman J, Bjorkelund C, Wallin L. Process evaluation of a cluster randomised intervention in Swedish primary care: using care managers in collaborative care to improve care quality for patients with depression. BMC Fam Pract. 2019 Jul 27;20(1):108. doi: 10.1186/s12875-019-0998-4. PMID 31351444